CLINICAL TRIAL: NCT05270577
Title: Pre-operative Prehabilitation in Cancer Surgery - Objective Recovery Assessment
Acronym: Popcorn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Bergthor Björnsson, Associate Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Popcorn
Record Dates: First submitted 2022-02-16; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Preoperative Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Prehabilitation with physical exercise, psychological support, nutritional support and smoking/alchohol stop
  Interventions: Other: Prehabilitation
- Standard care (Active Comparator): Standard preoperative recomendations
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Prehabilitation — prehabilitation
  Arms: Prehabilitation
Other: Standard care — No intervention
  Arms: Standard care

SUMMARY:
To compare prehabilitation with physical exercise, psychological support, nutritional support and smoke/alchol stop to "standard of care" before canceer surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients, aged 18 or older, who have been evaluated as eligible for surgery for malignancy in the esophagus, rectum or liver (only metastases from colorectal cancer) will be evaluated for participation.

Exclusion Criteria:

* Surgery is scheduled in less than 12 weeks.
* Paralytic or completely immobilized patient, condition making physical training impractical.
* Cognitive disability making participation impossible.
* Not speaking or understanding the Swedish language well enough to read and understand the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test (6mwt) | 12 weeks
  6 minute walk test (6mwt)

SECONDARY OUTCOMES:
30 s chair stand test | 12 weeks
  30 s chair stand test
Test of hand grip strength | 12 weeks
  Test of hand grip strength
International Physical Activity Questionnaire | 12 weeks
  International Physical Activity Questionnaire
Cardiopulmonary exercise test with ventilatory gas analysis | 12 weeks
  Cardiopulmonary exercise test with ventilatory gas analysis making it possible to calculate VOmax as well as other established measures of cardiopulmonary function
The presence of malnutrition evaluated with the Global Leadership Initiative on Malnutrition (GLM) criteria | 12 weeks
  The presence of malnutrition evaluated with the Global Leadership Initiative on Malnutrition (GLM) criteria
Appetite and eating behavior is evaluated with Eating Symptom Questionnaire (ESQ) | 12 weeks
  Appetite and eating behavior is evaluated with Eating Symptom Questionnaire (ESQ)
Appetite and eating behavior is evaluated with Disease Related Appetite Questionnaire (DRAQ) | 12 weeks
  Appetite and eating behavior is evaluated with Disease Related Appetite Questionnaire (DRAQ)
4-week point prevalence of smoking abstinence (among baseline smokers) | 12 weeks
  4-week point prevalence of smoking abstinence (among baseline smokers), measured with Fagerstroms scale
Weekly alcohol consumption | 12 weeks
  Weekly alcohol consumption as reported in standard units
Episodes of heavy drinking per month | 12 weeks
  Episodes of heavy drinking per month as reported in standard units at a single occation
The most severe complication occurring | 90d after surgery
  The most severe complication occurring (according to the Clavien-Dindo scale) until 90 days after surgery
Sum of all complications in each patient (comprehensive complication index, CCI) | 90d after surgery
  Sum of all complications in each patient (comprehensive complication index, CCI) occuring up to 90 days after surgery
Length of hospitalization | 90d after surgery
  Length of hospitalization
Time to functional recovery of physical status as compared to baseline values | 90d after surgery
  Defined as number of days after surgery until the patient has reached all of the following: being mobile at the preoperative level, having sufficient pain control with only oral or transdermal medication, being able to maintain food intake without intravenous fluids and not being in need of intravenous medications
Clinical Frailty Scale | 12 weeks
  Clinical Frailty Scale
Grade of sarcopenia | 12 weeks
  Grade of sarcopenia
The frequency of failures to go through the full treatment program as planned at the first MDT (including, but not limited to, the full oncological chemotherapy program, radiation treatment and final surgery) | 90 days
  The frequency of failures to go through the full treatment program as planned at the first MDT (including, but not limited to, the full oncological chemotherapy program, radiation treatment and final surgery)
Time from surgery until the day of first dose of adjuvant chemotherapy (among liver and rectal cancer patients for whom postoperative chemotherapy is planned) | 90 day after surgery
  Time from surgery until the day of first dose of adjuvant chemotherapy (among liver and rectal cancer patients for whom postoperative chemotherapy is planned)
Proportion of patients not able to receive all treatment despite no dissemination of disease | 90 day after surgery
  Proportion of patients not able to receive all treatment despite no dissemination of disease
Overall survival | 5 years
  Overall survival
Quality of Life (QoL) | 2 years after surgery
  Quality of Life (QoL)
Incremental cost-effectiveness ratio | 2 years after surgery
  Incremental cost-effectiveness ratio, calculated as the median cost divided by the quality adjusted life years obtained until 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bergthor Björnsson, MD, PhD, Principal Investigator — Linkoeping University

IPD SHARING:
Plan to Share IPD: No